CLINICAL TRIAL: NCT01178567
Title: Comparison of Pulmonary Complications Related to Laparoscopic Sleeve Gastrectomy and Laparoscopic Adjustable Gastric Banding
Brief Title: Comparison of Pulmonary Complications Related to Sleeve Gastrectomy and Gastric Banding
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10-117-10.CTIL
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: "Pulmonary Complications"
Keywords: laparoscopic sleeve gastrectomy; Gastrectomy; Pulmonary Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of Pulmonary Complications related to laparoscopic sleeve gastrectomy and laparoscopic adjustable gastric banding.

DETAILED DESCRIPTION:
Obesity is defined as a body mass index (BMI) of more than 30 (1). Its frequency varies according to social, economical and cultural situations. Approximately 15%-20% of the population of Europe, 40% of the United States, and up to 80% of some Native American and Pacific Islands populations (1) are morbidly obese, defined as a BMI more than 39 (2).

The laparoscopic adjustable silicone banding (LAP-BAND) procedure has rapidly gained acceptance and is now considered the most common bariatric operation. In the literature, there are rare case reports about respiratory complications following LAP-BAND. Hofer et al. (3) reported a case of recurrent aspiration pneumonia. Nemni reported a case of chronic cough that was eliminated after LAP-BAND deflation (4). Almoudi reported a case of left lower lobe pneumonia 3 years following LAP-BAND. The patient had presented with asthma-like symptoms (5).

However, there are no studies in the literature addressing long-term pulmonary complications following LAP-BAND. Reports on most previous studies with a medium-term follow-up of 4 years have focused on weight loss as a deciding factor for the success of the surgery, rather than on long-term complications.

Laparoscopic sleeve gastrectomy (LSG) is an innovative approach to the surgical management of morbid obesity (6). Early data suggest LSG is efficacious in the management of morbid obesity and may have an important role either as a staged or definitive procedure. A systematic review of the literature analyzing the clinical and operational outcomes of LSG was completed to further define the status of LSG as an emerging treatment modality for morbid obesity (7). Data from LSG were compared to benchmark clinical data and local operational data from laparoscopic adjustable gastric band (LAP-BAND) and laparoscopic gastric bypass (LRYGB) procedures.

A systematic review of the literature identified 15 studies (940 patients). The percent excessive weight loss (%EWL) for LSG varied from 33% to 90% and appeared to be sustained up to 3 years. The mortality rate was 0-3.3% and major complications ranged from 0% to 29% (average 12.1%). Operative time ranged from 49 to 143 min (average 100.4 min). Hospital stay varied from 1.9 to 8 days (average 4.4 days).

The operational impact of LSG has not been described in the literature. Early, non-randomized data suggest that LSG is efficacious in the surgical management of morbid obesity (8). However, it is not clear if weight loss following LSG is sustained long term and therefore, it is not possible to determine what percentage of patients may require additional revisional surgery following LSG. The operational impact of LSG as a staged or definitive procedure is poorly defined and must be analyzed further to establish its overall health care costs and operational impact. Although LSG is a promising treatment option for patients with morbid obesity, its role remains undefined and it should be considered an investigational procedure that may require revision in a subset of patients (9).

Although previous studies reported that both LSG and LAP-BAND resulted in postoperative improvement or resolution of comorbid conditions associated with obesity, LSG statistically showed a significantly higher rate of resolution or improvement of DM, HTN, and LPD. There was no significant difference between the groups for DJD, GERD, OSA, or asthma (2). The incidence of pulmonary complications was not reported.

This study will retrospectively compare the rates of pulmonary complications following LAP-BAND and LSG surgeries. The effect of the surgery on the comorbid conditions of type 2 diabetes mellitus (DM), hypertension (HTN), hyperlipidemia (LPD), degenerative joint disease (DJD), gastroesophageal reflux disease (GERD), obstructive sleep apnea (OSA), and asthma in the two subpopulations will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who paste surgery in Meir Hospital included with stomach ring and sleeve surgery.

Exclusion Criteria:

* Patients who underwent other bariatric surgery in the past will excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 sleeve gastectomy patients
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Comparison of Pulmonary Complications related to laparoscopic sleeve gastrectomy and laparoscopic adjustable gastric banding. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir MC, Kfar Saba, Israel, Israel